CLINICAL TRIAL: NCT07075783
Title: Comparison of Efficacy of MgSO4 Added to Ropivacaine and Ropivacaine Alone in Scalp Block for Craniotomy: a Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Magnesium Sulphate Adjuvant in Scalp Block With Ropivacaine for Supratentorial Craniotomy: a Prospective, Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Alwyn Lee Chee Yuan, Principal Investigator, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23110854
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Efficacy and Safety of MgSO4 as Adjuvant to Scalp Block
Keywords: Magnesium; MgSO4; Scalp block; Craniotomy; Supratentorial; Ropivacaine; Remifentanil; Adjuvant; Efficacy
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (RN) (Placebo Comparator): •Control (RN) group: 0.375% Plain Ropivacaine at a maximum recommended dose of 3 mg/kg body weight, plus 5 mcg/ml adrenaline and 1 ml of 0.9% NaCl.
  Interventions: Other: Plain Ropivacaine
- Study group (RM) (Experimental): Study (RM) group: 0.375% Plain Ropivacaine at maximum recommended dose of 3 mg/kg body weight, plus 5 mcg/ml adrenaline and 1 ml of 50% MgSo4.
  Interventions: Drug: MgSO4 plus Ropivacaine

INTERVENTIONS:
Drug: MgSO4 plus Ropivacaine — 1ml 50% MgSO4 added to 0.375% Plain Ropivacaine plus 5 mcg/ml adrenaline for scalp block
  Arms: Study group (RM)
Other: Plain Ropivacaine — 0.375% Plain Ropivacaine plus 5 mcg/ml adrenaline and 1 ml of 0.9% NaCl
  Arms: Control group (RN)

SUMMARY:
A randomized, double-blinded controlled trial was conducted to evaluate the analgesic efficacy of MgSO4 as an adjuvant to ropivacaine in scalp blocks for craniotomy, focusing on its impact on hemodynamic parameters and intraoperative remifentanil consumption.

DETAILED DESCRIPTION:
A prospective, randomized, double-blinded controlled trial was conducted at Hospital Universiti Sains Malaysia (HUSM). Twenty-four patients scheduled for elective supratentorial craniotomy under general anesthesia were randomized into two groups: the control group (ropivacaine alone) and the treatment group (ropivacaine with MgSO4). Hemodynamic parameters, including mean arterial pressure (MAP) and heart rate (HR), were recorded at seven predefined intraoperative time points corresponding to critical surgical stimuli. Total intraoperative remifentanil consumption was also measured.

ELIGIBILITY:
Inclusion Criteria:

* 1. Scheduled for elective supratentorial craniotomy under general anaesthesia 2. ASA I-III physical status 3. Aged 18 years and above

Exclusion Criteria:

* 1. Traumatic brain injury 2. Aneurysmal clipping 3. GCS <14 4. Contraindication to scalp block 5. Known adverse reaction to magnesium sulphate or LA from previous exposure 6. Heart block 7. History of drug dependence or alcohol abuse 8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Pressure | Mean arterial blood pressure (MAP) recorded at seven time points: scalp block (T0), skull pin fixation (T1), skin incision (T2), craniotomy (T3), durotomy (T4), dura mater closure (T5) and skin closure (T6)
Heart Rate (HR) | Heart Rate (HR) recorded at seven time points: scalp block (T0), skull pin fixation (T1), skin incision (T2), craniotomy (T3), durotomy (T4), dura mater closure (T5) and skin closure (T6)

SECONDARY OUTCOMES:
Cumulative remifentanil dose | Total intra-operative consumption of remifentanil

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided